CLINICAL TRIAL: NCT00297245
Title: Gastrodin Prevents Cognitive Decline Related to Cardiopulmonary Bypass
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 21124941
Record Dates: First submitted 2006-02-27; First posted 2006-02-28 (Estimated); Last update posted 2006-02-28 (Estimated); Status verified 2006-01

CONDITIONS: Cognitive Decline
Keywords: gastrodin
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Neuropsychological Tests

INTERVENTIONS:
Drug: cognitive function

SUMMARY:
The incidence of cognitive decline related to CPB ranges from 20% to 80%, which may affect length of hospital stay, quality of life, the rehabilitation process, and work performance.However, there is no method to prevent the decline.Gastrodin,the active constituent of gastrodia elata, has been widely used for the treatment of paralysis, hemiplegia, headache, vertigo, and Alzheimer's disease. Gastrodin is safe. No severe side-effect has been observed in the treatment. We postulate that gastrodin would attenuate the causative parameters of cognitive dysfunction related to CPB and would be an effective drug to prevent the decline as a result.

DETAILED DESCRIPTION:
Cardiac surgery with cardiopulmonary bypass (CPB) is one of the most frequently performed operations. Neurobehavioral disorders, including neuropsychiatric and neuropsychological deficits, are a very frequently reported sequela of valve replacement or coronary artery bypass grafting (CABG) surgery. CPB is associated with significant cerebral morbidity. The incidence of cognitive decline related to CPB ranges from 20% to 80%, which may affect length of hospital stay, quality of life, the rehabilitation process, and work performance. Neurocognitive decline can present days to weeks after surgery and may remain a permanent disorder. Many pharmacologic strategies have been proposed or investigated for preventing post-CPB cognitive decline, but to our knowledge, none of these drugs has been systematically evaluated for efficacy in preventing post-CPB cognitive decline.

The causative parameters of cognitive dysfunction associated with CPB include cerebral ischemia secondary to either microemboli or hypoperfusion, intraoperative cerebrovascular risk factors such as the duration of CPB, inflammatory response, cerebral glutamine release, free radicals, and NO release.

Gastrodia elata, a famous Chinese medical herb, has effects on preventing ischemic brain injury, neuronal cell damage or apoptosis, suppressing inflammatory response, inhibiting glutamine receptors and nNOS, and scavenging free radicals. Gastrodin (4-[hydroxymethyl]phenyl-β-D-glucopyranoside), the primary active constituent of gastrodia elata, has been widely used for the treatment of paralysis, hemiplegia, headache, vertigo, and Alzheimer's disease. Based on its pharmacological effects, we postulated that gastrodin would attenuate the causative parameters of cognitive dysfunction related to CPB and would be an effective drug to prevent the decline as a result.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergo mitral valve replacement surgery.

Exclusion Criteria:

* Thrombi in left atrium, a history of symptomatic cerebrovascular disease, diabetes, psychiatric illness, renal disease, or active liver disease, less than a seven-grade education, or who cannot read.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2006-02; Study Completion 2006-05

PRIMARY OUTCOMES:
Gastrodin markedly prevents cognitive decline related to cardiopulmonary bypass

SECONDARY OUTCOMES:
neuropsychological tests

CONTACTS AND LOCATIONS:
Overall Officials: Shihai Zhang, Principal Investigator — Department of Anesthesiology, Union Hosiptal, Tongji Medical College, Huazhong University of Science and Technology; Shihai Zhang, M.D., Ph.D., Principal Investigator — Department of Anesthesiology, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Department of Anesthesiology, Union Hospital, Wuhan, Hubei, China